CLINICAL TRIAL: NCT05916352
Title: The Effect of Caffeine Supplementation on Blood Lactate Level, Performance and Post-Training Fatigue in Elite Basketball Players
Brief Title: Effects of Caffeine on Upper Extremity Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sıddıka Fatma Uygur, Academic Professor, Cyprus International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: -020-7249
Record Dates: First submitted 2023-06-07; First posted 2023-06-23 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Sportive Performance; Caffeine
Keywords: Caffeine; Performance; Lactic Acid; Basketball; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: The research is a double-blind randomized controlled comparative cross-sectional study.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine Group (Active Comparator): 5 mg/kg caffein supplement will be given
  Interventions: Dietary Supplement: Caffeine Supplement
- Placebo Group (Placebo Comparator): Placebo will be given
  Interventions: Dietary Supplement: Caffeine Supplement

INTERVENTIONS:
Dietary Supplement: Caffeine Supplement — Caffeine tablet

SUMMARY:
It was aimed to apply caffeine supplement to elite basketball players and to investigate the effects of this supplement on upper extremity performance, lactic acid level and fatigue. The investigators also aimed to investigate the effects of blood lactate level on performance and fatigue.

DETAILED DESCRIPTION:
The aim of this study is to examine the effects of caffeine supplementation on upper extremity performance, lactic acid and fatigue in elite basketball players and compare them with the placebo group. A total of 50 elite basketball players, 25 each in the caffeine and placebo groups, will participate in the study. Caffeine supplement will be given 1 hour before the measurements (5mg/kg). Muscular endurance before and after reinforcement, scapular muscular endurance test (SKET); arm movement speed, disc touch test (DDT); anaerobic power, medicine ball throwing (STF); lactic acid (LA) level will be evaluated by finger blood measurement and fatigue visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Elite basketball players aged 19-44
* Individuals with caffeine consumption below 2 mg per kg per day

Exclusion Criteria:

* Individuals with systemic disease affecting the musculoskeletal system
* Individuals using supplements containing caffeine
* Individuals with any diagnosed neurological or orthopedic disease

Ages: 19 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Blood Lactate Level | 2 hours
  Lactic acid level in the blood

SECONDARY OUTCOMES:
Reaction Time | 5 minutes
  Arm movement speed
Anaerobic Power | 5 minutes
  Upper extremity explosive force will be measured with medicine ball
Muscular Endurance | 5 minutes
  Endurance time will be measured using a 1 kg Dynamometer.
Fatigue | 1 minute
  Subjective fatigue will be measured using the Visual Analog Scale which ranging from 0 to 10 points. A value of 0 describes "no pain" and a value of 10 describes the "most pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Cyprus International University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data obtained from the participants will be shared in the form of thesis and scientific articles.
Supporting Information: Study Protocol
Time Frame: Starting in July 2023
Access Criteria: The results of the study will be shared in the form of scientific articles by making appropriate statistical analyzes.

REFERENCES:
- [Result] Ben Abdelkrim N, Castagna C, El Fazaa S, Tabka Z, El Ati J. Blood metabolites during basketball competitions. J Strength Cond Res. 2009 May;23(3):765-73. doi: 10.1519/JSC.0b013e3181a2d8fc. PMID 19387403
- [Result] Spriet LL. Exercise and sport performance with low doses of caffeine. Sports Med. 2014 Nov;44 Suppl 2(Suppl 2):S175-84. doi: 10.1007/s40279-014-0257-8. PMID 25355191
- [Result] Burke LM. Practical Issues in Evidence-Based Use of Performance Supplements: Supplement Interactions, Repeated Use and Individual Responses. Sports Med. 2017 Mar;47(Suppl 1):79-100. doi: 10.1007/s40279-017-0687-1. PMID 28332111
- [Result] Caravan I, Sevastre Berghian A, Moldovan R, Decea N, Orasan R, Filip GA. Modulatory effects of caffeine on oxidative stress and anxiety-like behavior in ovariectomized rats. Can J Physiol Pharmacol. 2016 Sep;94(9):961-72. doi: 10.1139/cjpp-2015-0502. Epub 2016 Apr 16. PMID 27333093
- [Result] Chia JS, Barrett LA, Chow JY, Burns SF. Effects of Caffeine Supplementation on Performance in Ball Games. Sports Med. 2017 Dec;47(12):2453-2471. doi: 10.1007/s40279-017-0763-6. PMID 28741186
- [Result] Grgic J, Trexler ET, Lazinica B, Pedisic Z. Effects of caffeine intake on muscle strength and power: a systematic review and meta-analysis. J Int Soc Sports Nutr. 2018 Mar 5;15:11. doi: 10.1186/s12970-018-0216-0. eCollection 2018. PMID 29527137
- [Result] Sant'Ana J, Franchini E, da Silva V, Diefenthaeler F. Effect of fatigue on reaction time, response time, performance time, and kick impact in taekwondo roundhouse kick. Sports Biomech. 2017 Jun;16(2):201-209. doi: 10.1080/14763141.2016.1217347. Epub 2016 Sep 5. PMID 27592682
- [Result] San Juan AF, Lopez-Samanes A, Jodra P, Valenzuela PL, Rueda J, Veiga-Herreros P, Perez-Lopez A, Dominguez R. Caffeine Supplementation Improves Anaerobic Performance and Neuromuscular Efficiency and Fatigue in Olympic-Level Boxers. Nutrients. 2019 Sep 5;11(9):2120. doi: 10.3390/nu11092120. PMID 31492050